CLINICAL TRIAL: NCT03798210
Title: The Effect of Lactobacillus Reuteri ATCC PTA 4659 in Patients With Ulcerative Colitis
Brief Title: Lactobacillus Reuteri ATCC PTA 4659 in Ulcerative Colitis
Acronym: COLUS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Uppsala University (Other)
Responsible Party: Principal Investigator, Per Hellström, Prof, MD, PhD, Uppsala University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: ATCC PTA 4659
Record Dates: First submitted 2019-01-07; First posted 2019-01-09 (Actual); Last update posted 2019-01-14 (Actual); Status verified 2019-01

CONDITIONS: Ulcerative Colitis Flare
Keywords: ulcerative colitis; prevention; microbiota; Lactobacillus
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Intervention Model Description: Lactobacillus reuteri versus placebo on prevention of flare in ulcerative colitis/proctosgmoiditis
Who Masked: Participant, Care Provider, Investigator
Masking Description: Pre-masked randomized tablet vials with Lactobacillus reuteri, or corresponding placebo
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Look and taste-alike placebo tablets in white plastic vials.
  Interventions: Dietary Supplement: Placebo
- Lactobacillus reuter's (Experimental): Lactobacillus reuteri tablets in white plastic vials.
  Interventions: Dietary Supplement: Lactobacillus reuteri

INTERVENTIONS:
Dietary Supplement: Lactobacillus reuteri — Study group split in two arms for experimental treatment with Lactobacillus reuteri or placebo.
  Arms: Lactobacillus reuter's
Dietary Supplement: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Explorative investigation to study the effect of the endogenous bacterium Lactobacillus reuteri ATCC PTA 4659 as a nutrient additive against relapse in ulcerative colitis. Forty patients will be studied with a randomized parallel design over one year. Patients with established treatment against relapse of ulcerative colitis with mesalazine ≤4 grams will be requested to participate in the study, allocated to 20 patients with placebo and 20 with active treatment L. reuteri as an "add-on". Inklusion: 18-80 years of age, ≥1 relapse with bleeding during previous 12 months with a disease activity Mayo Clinical Score ≤2, treatment with mesalazine ≤4,0 g daily. Exklusion: >80 years of age, no registered bleeding during recent 12 months, on-going steroid treatment, immunosuppressives, biologics or adhesion inhibitors, antibiotics or other clinical trial. behandling med probiotika. Disease monitoring will be done with:

Time to disease relapse with macroscopic bleeding and Mayo score ≥5, blood chemistry and CRP, lipopolysaccharides and gut permeability, fecal calprotectin, and short health scale at 4 weeks, 26 weeks and 52 weeks.

DETAILED DESCRIPTION:
Research question To study whether dietary supplementation with L. reuteri ATCC PTA 4659 (Lr4659) is safe and can reduce the relapse rate and have a positive effect in patients with ulcerative colitis (UC).

Lr4659 is a naturally occurring strain of human origin. It is a typical member of the L. reuteri species, with typical sugar fermentation patterns, reuterin production and growth characteristics. Identification using 16SrRNA gene analysis shows that it has 99% similarity with the type strain of L. reuteri thus confirming that it belongs to this well-known and well-studied species that is considered safe for human consumption. In vitro studies indicate that this strain has strong tolerance to acid environments, as do many other L. reuteri strains and that it has the unusual ability to interfere with TNFalpha mediated propagation of inflammatory responses in human macrophages.

Treatment with the probiotic bacterium L. reuteri has been shown to prevent dextran sodium sulfate (DSS)-induced colitis in rats. During DSS-induced colitis, the number of bacteria in the inner firmly-adherent mucus layer increased and bacterial composition of the two layers no longer differed. However, L. reuteri decreased the bacterial translocation from the intestine to mesenteric lymph nodes during DSS treatment, which might be an important part of the mechanisms by which L. reuteri ameliorates DSS-induced colitis in rats.

Study design This is a double-blind randomized clinical trial. Randomization will be done to either mesalazine plus Lr4659, or to mesalazine plus placebo for a continuous treatment until new bleeding episode or a maximum of 52 weeks.

Forty patients with UC in remission, medicated with <4 g mesalazine and aged over 18 years will be recruited. After written consent to the study the subjects in whom the eligibility criteria are confirmed the subjects will be randomized to receive either 2 daily doses of Lr4659 (n=15) or the corresponding placebo. The total length of study treatment is 52 weeks.

Concomitant treatment During the period of the study, the subjects will refrain from ingestion of any kind of probiotic or bacterial preparation.

The objective is to determine whether dietary supplementation with Lr4659 is able to: Prolong time in remission and Time from last bleeding episode until re-bleeding, Time from start of study treatment until re-bleeding, Reduce Mayo score reduction by at least 50%, Reduce f-calprotectin, Reduce recovered sucralose in the sucralose gut permeability test, Reduce zonulin expression from gut mucosa, Impact microflora composition

Study Product and Dosage Lr4659, consisting of L. reuteri ATCC PTA 4659 will be delivered at a dose of 5x108 colony forming units (CFU) as a powder in capsules. One dose is to be taken in the morning and one in the evening yielding a total daily dose of 1x109 CFU/day. Placebo capsules are identical to Lr4659 except for the active ingredient. The study products will be taken daily throughout the entire 52-week study-period.

Inclusion criteria for study: UC confirmed by biopsy, Mayo full score < 2, Total or left-sided UC, Stable diagnose of UC >1 year, History of more than 1 yearly recurrence, Current remission period exceeding 2 months, 18-80 years of age, Baseline 5-ASA ≤4g daily, Mentally fit to participate, Informed consent obtained Exclusion criteria: Crohn's disease, Ulcerative proctitis, Infective colitis, Liver disease, Current use of probiotics, Current medication acetylsalicylic acid (ASA), non-steroidal antiinflammatory drugs (NSAID), corticosteroids, anticoagulants, serotonin-selective re-uptake inhibitors (SSRI), serotonin-noradrenaline re-uptake inhibitors (SNRI), azathioprine (AZA), 6-mercaptopurin (6-MP), thioguanin (TG), anti-TNF-alpha biologicals, Participation in other clinical trials

Analyses Evaluation of the clinical Mayo score will be done by ocular inspection and immediate recording in the CRF.

C-reactive protein (CRP) will be locally analysed according to clinical routine by Department of clinical chemistry, Uppsala University Hospital.

Fecal calprotectin will be analysed according to local routines (Bühlmann, Schönenbuch, Switzerland) by Department of clinical chemistry, Uppsala University Hospital).

"Gut" permeability focuses on colonic permeability as studied with recovery of different sugar components in the urine. 24-hour urine will be analysed by an in-house high performance liquid chromatography (HPLC) method by GastroLab, Uppsala University Hospital.

Fecal microbiology, alfa-diversity, beta-diversity

Expected findings: Prolonged interval to next flare of UC with rectal bleeding. Reduced calprotectin and CRP levels.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of UC confirmed by biopsy
* Mayo full score < 2
* Total or left-sided UC
* Stable diagnose of UC >1 year
* History of more than 1 yearly recurrence
* Current remission period exceeding 2 months
* 18-75 years of age
* Baseline 5-ASA ≤2g daily
* Mentally fit to participate
* Informed consent obtained

Exclusion Criteria:

* Crohn's disease
* Ulcerative proctitis
* Infective colitis
* Liver disease
* Current use of probiotics
* Current medication acetylsalicylic acid (ASA), non-steroidal antiinflammatory drugs (NSAID), corticosteroids, anticoagulants, serotonin-selective re-uptake inhibitors (SSRI), serotonin-noradrenaline re-uptake inhibitors (SNRI), azathioprine (AZA), 6-mercaptopurin (6-MP), thioguanin (TG), anti-TNF-alpha biologicals
* Participation in other clinical trials

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-01-31 (Estimated); Study Completion 2019-03-01 (Estimated)

PRIMARY OUTCOMES:
Rectal bleeding with Mayo score ≥5 | 12 months
  Rectal bleeding as sign of increased inflammatory activity as determined by the Mayor Clinic Score for evaluation of disease activity in ulcerative colitis

SECONDARY OUTCOMES:
Increased fecal calprotectin | 12 months
  Gut inflammatory biomarker
Increased CRP | 12 months
  General inflammatory biomarker

OTHER OUTCOMES:
Serum Zonulin | 12 months
  Gut permeability biomarker
Gut permeability | 12 months
  Recovery of sugar molecules in urine as marker of increased permeability

CONTACTS AND LOCATIONS:
Overall Officials: Per M Hellström, Prof, Principal Investigator — Uppsala University
Locations (1):
- Uppsala University, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: Undecided
Shared at publication.